CLINICAL TRIAL: NCT05340842
Title: Evaluation of the Effects of Simulation Based Breastfeeding Training on Women' Breastfeeding Success, Breastfeeding Self Efficacy, Breastfeeding Attitude and Knowledge
Brief Title: Evaluation of the Effects of Simulation Based Breastfeeding Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Hamide Aslan, Research Assistant, Principal Investigator, Marmara University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16214662/050.01.04/30
Record Dates: First submitted 2022-04-04; First posted 2022-04-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Breastfeeding; Education
Keywords: antenatal period; simulation based breastfeeding training
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation training experiment group (Experimental): In this training, the researcher firstly explained breastfeeding by wearing the Lactation Simulation Model on himself and showing it practically on himself.
  Afterwards, the model was dressed on the pregnant woman and the pregnant woman was given one-on-one breastfeeding practice.
  In this process, all questions of the pregnant woman were answered by the researcher.
  Interventions: Other: simulation training group
- Control group (No Intervention): At this stage, the standard video screening prepared for breastfeeding education within the scope of the hospital protocol was shown to the pregnant woman by the researcher with a tablet.

INTERVENTIONS:
Other: simulation training group — In this study, applied breastfeeding training with Lactation Simulation Model was given to pregnant women in the intervention group (simulation training group, n=64) during antenatal period
  Arms: Simulation training experiment group

SUMMARY:
This study is a randomized controlled experimental study conducted to determine the effect of applied breastfeeding training given through Lactation Simulation Model (LSM) in antenatal period on the success of women in breastfeeding, their self-efficacy perception regarding breastfeeding and their attitude towards and knowledge of breastfeeding.

DETAILED DESCRIPTION:
This study is a randomized controlled experimental study conducted to determine the effect of applied breastfeeding training given through Lactation Simulation Model (LSM) in antenatal period on the success of women in breastfeeding, their self-efficacy perception regarding breastfeeding and their attitude towards and knowledge of breastfeeding. The research was carried out with the participation of two groups. In this context, applied breastfeeding training with LSM was given to pregnant women in the intervention group (simulation training group, n=64) during antenatal period, and standard training-video training under the hospital protocol (video training group, n = 64) was provided to pregnant women in the control group. Then, breastfeeding success, breastfeeding self efficacy, attitude and knowledge levels regarding breastfeeding were evaluated in the postnatal period. The data of the research were collected through Participant Description Questionnaire, LATCH Assessment Tool, Breastfeeding Attitude and Knowledge Questionnaire, Breastfeeding Self efﬁcacy Scale and Postnatal Period Follow-up Questionnaire. In addition, LSM was employed in the implementation for the simulation training group. Research data were analyzed by using SPSS 23.0 statistics program.

ELIGIBILITY:
Inclusion Criteria:

32-36 between gestational weeks Primigravida No systemic/chronic disease Planning to breastfeed Who has not received a planned breastfeeding training before Can speak and understand Turkish Pregnant women who agreed to participate in the study were included.

Exclusion Criteria:

Breastfeeding contraindications Having a high-risk pregnancy Preterm delivery (before 37 weeks of gestation) Having a health condition that prevents breastfeeding in the newborn after birth Having mental disability and serious mental disorder Women with multiple pregnancies were excluded from the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
LATCH Breastfeeding Diagnostic and Assessment Scale | The scale was filled twice, with an average of two hours, in the first 24 hours after delivery, when the mother was free of pain and felt well.
  LATCH consists of the combination of the first letters of the English equivalent of the five criteria defined above. Each item is evaluated between 0-2 points. The lowest score that can be obtained from the entire scale is 0 and the highest score is 10. The scale has no breakpoints. The low score on the scale indicates the need for active intervention, support and follow-up after discharge in breastfeeding. The higher the LATCH Breastfeeding Diagnosis and Evaluation Scale score, the higher the success of breastfeeding. Cronbach's alpha value was found to be 0.95 in the study in which the Turkish validity and reliability of the scale was carried out.

SECONDARY OUTCOMES:
Breastfeeding Attitude and Knowledge Questionnaire | It was applied both in the antenatal period (at 32-36 weeks of pregnancy) and in the postnatal 24 hours.
  This form was created by researchers in line with the literature in order to determine the attitudes and knowledge levels of pregnant women towards breastfeeding.In the form, there are a total of 20 statements, 10 statements questioning the level of knowledge about breastfeeding and 10 statements questioning the attitude towards breastfeeding. Each statement in the form is marked as "True", "Wrong", "I don't know" according to the attitude and knowledge level of the people. In the evaluation of the form, correct answers were given as "1", "I don't know" or wrong answers were given "0" points. The lowest score that can be obtained from the entire form is 0 and the highest score is 20. The Cronbach's alpha value of the attitude and knowledge evaluation form regarding breastfeeding was found to be 0.60 in the antenatal period and 0.75 in the postnatal period. A high score on the form indicates a high level of positive attitude and knowledge about breastfeeding.
Breastfeeding Self-Efficacy Scale-Short Form | It was applied both in the antenatal period (at 32-36 weeks of pregnancy) and in the postnatal 24 hours.
  Breastfeeding Self-Efficacy Scale consists of 14 items. The lowest score that can be obtained from the entire scale is 14 and the highest score is 70. A high score from the scale indicates a high perception of breastfeeding self-efficacy. This scale can be applied both in the antenatal and postnatal periods. The difference of the antenatal form of the scale from the postnatal form is that the phrase "future tense" is used in the scale items. In the original study of the scale, the Cronbach's alpha value of the antenatal form was 0.87, and the Cronbach's alpha value of the postnatal form was 0.86.

CONTACTS AND LOCATIONS:
Overall Officials: Hamide Arslan Tarus, Res. Asist., Principal Investigator — Marmara University; Gonul Kurt, Assist. Prof, Study Director — Gulhane Faculty of Nursing
Locations (1):
- Hamide Arslan Tarus, Istanbul, Maltepe, Turkey (Türkiye)